CLINICAL TRIAL: NCT01929746
Title: A Single-Dose, Single-Blind, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BIIB019, Daclizumab High Yield Process (DAC HYP), in Japanese and Caucasian Adult Healthy Volunteers
Brief Title: Daclizumab Japanese PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205HV102; EUDRA CT NO: 2013-002310-12
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — daclizumab HYP

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- BIIB019, 75 mg (Experimental): BIIB019 delivered via Subcutaneous Injection
  Interventions: Biological: BIIB019 subcutaneous injection
- BIIB019, 150 mg (Experimental): BIIB019 delivered via Subcutaneous Injection
  Interventions: Biological: BIIB019 subcutaneous injection

INTERVENTIONS:
Biological: BIIB019 subcutaneous injection — participants will be randomized to receive a single subcutaneous injection of BIIB019, 75 mg or 150 mg per dose group
  Other Names: Daclizumab High Yield Process; DAC HYP

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetic (PK) profile of BIIB019 (Daclizumab High Yield Process; DAC HYP) administered as a single subcutaneous (SC) dose (75 mg or 150 mg) Japanese and Caucasian adult healthy volunteers. The secondary objective of this study in this study population is to assess the safety and tolerability of BIIB019 administered as a single SC dose (75 mg or 150 mg).

ELIGIBILITY:
Key Inclusion Criteria:

* Japanese subjects must have been born in Japan, have both parents and grandparents of Japanese origin, and not have lived outside of Japan for more than 5 years or significantly modified their diets since leaving Japan.
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for at least 4 months after their last dose of study treatment.
* Body mass index (BMI) within 18 to 30 kg/m2, inclusive.
* Nonsmoker or be willing to abstain from using tobacco and tobacco-containing products for 24 hours prior to clinic admission and during the In-Clinic Period and to smoke no more than 10 cigarettes per day throughout the remainder of the study.
* Must be willing to refrain from all alcohol consumption for 48 hours prior to Day 1 and during the In-Clinic Period and to limit the intake of alcohol to no more than 2 units per day throughout the remainder of the study.

Key Exclusion Criteria:

* History of a positive test result for human immunodeficiency virus (HIV) antibody.
* History of hepatitis or a positive test result for hepatitis C virus antibody (HCVAb) or hepatitis B virus antibody (test for hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb]).
* History of tuberculosis (TB) or a positive QuantiFERON®-TB Gold test. There must be no other clinical evidence of TB on physical examination of the subject. Note: Subjects who have had prior adequate prophylaxis treatment for latent TB with an appropriate course of isoniazid or equivalent, per country standards, are not excluded from study participation.
* Subjects with a history of carcinoma in situ and malignant disease, with the exception of basal cell carcinoma that has been completely excised prior to study, are not eligible.
* Treatment with any prescription medication within 2 weeks before Day -1 with the exception of oral contraceptives for women of childbearing potential.
* Treatment with any nonprescription medicinal products (including vitamin/mineral/herbal-containing preparations but excluding acetaminophen) within the 7 days prior to study treatment.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUCinf) | Up to Day 105
Maximum observed concentration (Cmax) | Up to Day 105
Time to reach maximum observed concentration (Tmax) | Up to Day 105
Terminal elimination half-life (t1/2) | Up to Day 105
Apparent volume of distribution (Vd/F) | Up to Day 105
Apparent clearance (CL/F) | Up to Day 105

SECONDARY OUTCOMES:
The number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 105

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Leeds, United Kingdom